CLINICAL TRIAL: NCT07098156
Title: Neuroanatomical Differences Associated With Anorexia Nervosa and Masking Behaviour in Autistic Individuals
Brief Title: Neural Correlates of Autistic Individuals With Anorexia Nervosa
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 349220
Record Dates: First submitted 2025-07-16; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Autism; Anorexia Nervosa
Keywords: MRI; Magnetic Resonance Imaging
MeSH Terms: conditions — Autistic Disorder; Anorexia Nervosa | interventions — Demography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autistic Control: Autistic individuals with no history of an eating disorder
  Interventions: Other: Single Research Visit 3T MRI Research Scan; Other: Demographic and Behavioural Questionnaires
- Autistic Patient: Autistic individuals acutely ill with anorexia nervosa
  Interventions: Other: Single Research Visit 3T MRI Research Scan; Other: Demographic and Behavioural Questionnaires

INTERVENTIONS:
Other: Single Research Visit 3T MRI Research Scan — Single research visit scan performed with a 3T magnetic resonance imaging scanner.
Other: Demographic and Behavioural Questionnaires — A series of demographic and behavioural questionnaires to be completed by participants, either online or during the single study visit. Questionnaires include the Eating Disorder Examination Questionnaire, Autism Spectrum Quotient, Monotropism Questionnaire, Camouflaging Autistic Traits Questionnaire, Hospital Anxiety and Depression Scale, Adult Attention Deficit Hyperactivity Disorder Self-Report Scale, Work and Social Adjustment Scale, International Trauma Questionnaire and Leibowitz Social Anxiety Scale. These questionnaires will also include a demographic questionnaire to acquire measures such as age, BMI, co-occurring conditions, etc.

SUMMARY:
Masking is a behaviour or strategy used by many Autistic people to appear non-Autistic and blend in with a neurotypical society. The goal of this observational study is to understand the relationship between masking, anorexia nervosa symptoms and brain structure in Autistic people. The main questions this study aims to answer are:

* Do Autistic individuals with anorexia nervosa show differences in structure or function of the brain relation to Autistic individuals without anorexia nervosa?
* Do Autistic individuals with anorexia nervosa display higher levels of masking than Autistic individuals without anorexia nervosa?
* Are there indeed relationships between levels of masking, anorexia nervosa symptoms and brain structure in Autistic people?

Researchers will compare Autistic people without anorexia nervosa to Autistic people with anorexia nervosa to see if there are differences between groups. Participants will:

* Complete a series of questionnaires focused on eating disorder symptoms, autistic traits, autistic masking and psychological well-being
* Undergo an MRI scan at the Aberdeen Royal Infirmary

DETAILED DESCRIPTION:
Autism is a neurodevelopmental condition and presents as a distinct neurotype, characterised by a wide range of social and behavioural differences, including divergences in cognitive thinking and methods of communication. Autism shares significant behavioural features with restrictive eating disorders (EDs) such as anorexia nervosa (AN). Those with AN exhibit significantly elevated levels of Autistic characteristics, ranging between 2%-53%. Importantly, a characteristic shown by some Autistic people is the presence of masking, a term describing a strategy used by Autistic people, whether conscious or unconscious, to 'blend in' with neurotypical peers. While initially overlooked, it is now well-known that masking behaviour can produce detrimental effects on Autistic individuals' mental health. The presence of masking behaviour has been associated with increased levels of physical and mental exhaustion, anxiety/depression, and importantly, an increased presence of EDs.

The Eating Disorder and Autism Collaborative (EDAC) used an arts-based method called Photovoice to capture the experiences of Autistic individuals with lived/living experience of an ED. Participants commented on the how an ED can serve as a means to mask or camouflage within a neurotypical world (e.g., an Autistic person may use restrictive eating or excessive exercise as a means with which to 'fit in' with their peers). Magnetic resonance imaging (MRI) research can assist in understanding which regions of the brain are associated with masking behaviour, and whether there are differences in brain function/structure in Autistic individuals with versus without an ED.

Structural magnetic resonance imaging (MRI) research reports similarities in brain structure between those with AN and Autistic individuals, reporting differential structure of the amygdala, cerebellum, insula, cingulate cortex, as well as orbitofrontal and frontal cortex in both groups. Shared differences extend to neuroanatomical parameters essential for brain development and connectivity, such as cortical thickness and surface area. Further, there are no studies investigation structural correlates with masking behaviour, or distinct aspects of social camouflage such as masking, assimilation and compensation. Further research is necessary to disentangle the complex relationship between Autistic characteristics and symptomatology associated with restrictive EDs.

The investigators believe that by further understanding the brain structure and function associated with ED symptomatology and masking behaviour in Autistic individuals can assist with the development of novel or tailored interventions for EDs in this community.

ELIGIBILITY:
Inclusion Criteria:

Healthy Autistic Individuals (Autistic Controls) must:

* Be aged 25-45 years
* Be Autistic (clinically diagnosed and/or have an Autism Quotient (AQ-10) score of ≥6)
* Be able to provide informed consent for the study
* Be able to read, understand and respond to questionnaires in English
* Have no history of an eating disorder
* Willing to have an MRI scan in Aberdeen

Autistic Individuals with anorexia nervosa must:

* Be aged 25-45 years
* Be Autistic (clinically diagnosed and/or have an AQ-10 score of ≥6)
* Be able to provide informed consent to the study
* Be able to read, understand and respond to questionnaires in English
* Have a diagnosis of anorexia nervosa or a body mass index of <18.5
* Willing to have an MRI scan in Aberdeen

Exclusion Criteria:

Individuals are not eligible for the study if they:

* Are aged <25 or >45 years
* Are not Autistic or not clinically diagnosed as Autistic and have an AQ-10 score of <6
* Are diagnosed with an eating disorder other than anorexia nervosa
* Have a history of brain injury (e.g., stroke)
* Be unable to provide informed consent for the study
* Have contraindications to MRI scanning, such has implantable cardiac devices
* Are unable to read, understand and respond to questionnaires in English
* As participants will need to consent to the study and complete questionnaires by themselves, individuals with intellectual disability will be excluded from this study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population for this study consists of Autistic individuals who both present or do not present with acute anorexia nervosa. Study population will be recruited from Scotland, primarily the NHS Grampian region.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Structural and Functional Brain Differences | From enrolment to single research visit (up to 30 weeks).
  To examine whether Autistic individuals with anorexia nervosa exhibit differences in brain structure or function relative to Autistic individuals without anorexia nervosa via 2-sample t-tests. Brain structure will be measured using surface and subcortical parcellations (in mm^3) acquired from Freesurfer. Brain functional connectivity at resting state will be measured using bivariate correlations of mean BOLD signal across pairs of regions of interest, converted to normally distributed scores using Fisher's transformation.
Levels of Masking | From enrolment to single research visit (up to 30 weeks).
  To determine whether Autistic individuals with anorexia nervosa exhibit higher masking behaviour than Autistic individuals without anorexia nervosa via 2-sample t-tests on total and subscale scores on the Camouflaging Autistic Traits Questionnaire. The Camouflaging Autistic Traits Questionnaire contains 25 statements relating to three subcategories of camouflaging (9 statements for the compensation subscale; 8 statements for the masking subscale; 8 statements for the assimilation subscale). All statements are scored on a scale of 1-7, and the scoring range on this measurement ranges from 25 to 175. Higher scores reflect greater camouflaging, with a threshold score of high camouflaging consisting of a score of 100 or greater.
Associations Between Masking, Anorexic Symptoms and Brain Structure | From enrolment to single research visit (up to 30 weeks).
  To determine if there are associations between the levels of masking, eating disorder symptomatology and brain structure in Autistic individuals via multiple 3-path mediation analysis established using generalised linear models.
  Levels of masking will comprise of total and scores on the Camouflaging Autistic Traits Questionnaire, which contains 25 statements. All statements are scored on a scale of 1-7, with a scoring range of 25-175. Higher scores reflect greater camouflaging, with a threshold score of consisting of 100 or greater.
  Levels of eating disorder symptomatology will comprise of the Eating Disorder Examination Questionnaire, which contains 28 statements. Total scores range from 0-6, with a clinical cut-off score of 2.8 for women, and 1.68 for men.
  Brain structure will be measured using surface and subcortical parcellations (in mm^3) acquired from Freesurfer.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Lilian Sutton Building, Aberdeen, Aberdeen City
  - NHS Grampian Eating Disorder Services, Aberdeen, Aberdeen City

IPD SHARING:
Plan to Share IPD: No
Our previous research with Autistic collaborators highlighted concerns regarding future use of their data for research that may harm Autistic identity. As such, IPD may only be available upon request from the principal investigators of this study and are subject to future ethical approval.

REFERENCES:
- [Background] Hull L, Mandy W, Lai MC, Baron-Cohen S, Allison C, Smith P, Petrides KV. Development and Validation of the Camouflaging Autistic Traits Questionnaire (CAT-Q). J Autism Dev Disord. 2019 Mar;49(3):819-833. doi: 10.1007/s10803-018-3792-6. PMID 30361940
- [Background] Leppanen J, Sedgewick F, Cardi V, Treasure J, Tchanturia K. Cortical morphometry in anorexia nervosa: An out-of-sample replication study. Eur Eat Disord Rev. 2019 Sep;27(5):507-520. doi: 10.1002/erv.2686. Epub 2019 Jun 6. PMID 31172616
- [Background] Nickel K, Joos A, Tebartz van Elst L, Matthis J, Holovics L, Endres D, Zeeck A, Hartmann A, Tuscher O, Maier S. Recovery of cortical volume and thickness after remission from acute anorexia nervosa. Int J Eat Disord. 2018 Sep;51(9):1056-1069. doi: 10.1002/eat.22918. Epub 2018 Sep 13. PMID 30212599
- [Background] Vijayakumar N, Allen NB, Youssef G, Dennison M, Yucel M, Simmons JG, Whittle S. Brain development during adolescence: A mixed-longitudinal investigation of cortical thickness, surface area, and volume. Hum Brain Mapp. 2016 Jun;37(6):2027-38. doi: 10.1002/hbm.23154. Epub 2016 Mar 4. PMID 26946457
- [Background] Sader M, Williams JHG, Waiter GD. A meta-analytic investigation of grey matter differences in anorexia nervosa and autism spectrum disorder. Eur Eat Disord Rev. 2022 Sep;30(5):560-579. doi: 10.1002/erv.2915. Epub 2022 May 7. PMID 35526083
- [Background] Alfano V, Mele G, Cotugno A, Longarzo M. Multimodal neuroimaging in anorexia nervosa. J Neurosci Res. 2020 Nov;98(11):2178-2207. doi: 10.1002/jnr.24674. Epub 2020 Aug 7. PMID 32770570
- [Background] Doyle-Thomas KA, Kushki A, Duerden EG, Taylor MJ, Lerch JP, Soorya LV, Wang AT, Fan J, Anagnostou E. The effect of diagnosis, age, and symptom severity on cortical surface area in the cingulate cortex and insula in autism spectrum disorders. J Child Neurol. 2013 Jun;28(6):732-9. doi: 10.1177/0883073812451496. Epub 2012 Jul 25. PMID 22832774
- [Background] Sydnor LM, Aldinger KA. Structure, Function, and Genetics of the Cerebellum in Autism. J Psychiatr Brain Sci. 2022;7:e220008. doi: 10.20900/jpbs.20220008. Epub 2022 Oct 25. PMID 36425354
- [Background] Fonville L, Giampietro V, Williams SC, Simmons A, Tchanturia K. Alterations in brain structure in adults with anorexia nervosa and the impact of illness duration. Psychol Med. 2014 Jul;44(9):1965-75. doi: 10.1017/S0033291713002389. Epub 2013 Sep 27. PMID 24074139
- [Background] Wronski ML, Geisler D, Bernardoni F, Seidel M, Bahnsen K, Doose A, Steinhauser JL, Gronow F, Boldt LV, Plessow F, Lawson EA, King JA, Roessner V, Ehrlich S. Differential alterations of amygdala nuclei volumes in acutely ill patients with anorexia nervosa and their associations with leptin levels. Psychol Med. 2023 Oct;53(13):6288-6303. doi: 10.1017/S0033291722003609. Epub 2022 Dec 5. PMID 36464660
- [Background] Schumann CM, Bauman MD, Amaral DG. Abnormal structure or function of the amygdala is a common component of neurodevelopmental disorders. Neuropsychologia. 2011 Mar;49(4):745-59. doi: 10.1016/j.neuropsychologia.2010.09.028. Epub 2010 Oct 13. PMID 20950634
- [Background] Duffy F, Gillespie-Smith K, Sharpe H, Buchan K, Nimbley E, Maloney E, Sader M, Kettley S, Kerr-Gaffney J, Waiter G, Tchanturia K. Eating Disorder and Autism Collaborative project outline: promoting eating disorder research embedded in a neurodiversity-affirming culture. BJPsych Bull. 2025 Aug;49(4):272-277. doi: 10.1192/bjb.2024.61. PMID 39113248
- [Background] Cassidy S, Bradley L, Shaw R, Baron-Cohen S. Risk markers for suicidality in autistic adults. Mol Autism. 2018 Jul 31;9:42. doi: 10.1186/s13229-018-0226-4. eCollection 2018. PMID 30083306
- [Background] Beck JS, Lundwall RA, Gabrielsen T, Cox JC, South M. Looking good but feeling bad: "Camouflaging" behaviors and mental health in women with autistic traits. Autism. 2020 May;24(4):809-821. doi: 10.1177/1362361320912147. PMID 32429817
- [Background] Bargiela S, Steward R, Mandy W. The Experiences of Late-diagnosed Women with Autism Spectrum Conditions: An Investigation of the Female Autism Phenotype. J Autism Dev Disord. 2016 Oct;46(10):3281-94. doi: 10.1007/s10803-016-2872-8. PMID 27457364
- [Background] Leppanen J, Sedgewick F, Halls D, Tchanturia K. Autism and anorexia nervosa: Longitudinal prediction of eating disorder outcomes. Front Psychiatry. 2022 Sep 21;13:985867. doi: 10.3389/fpsyt.2022.985867. eCollection 2022. PMID 36213911
- [Background] Nickel K, Maier S, Endres D, Joos A, Maier V, Tebartz van Elst L, Zeeck A. Systematic Review: Overlap Between Eating, Autism Spectrum, and Attention-Deficit/Hyperactivity Disorder. Front Psychiatry. 2019 Oct 10;10:708. doi: 10.3389/fpsyt.2019.00708. eCollection 2019. PMID 31649563
- [Background] Westwood H, Tchanturia K. Autism Spectrum Disorder in Anorexia Nervosa: An Updated Literature Review. Curr Psychiatry Rep. 2017 Jul;19(7):41. doi: 10.1007/s11920-017-0791-9. PMID 28540593
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders. 5th ed. Arlington, VA: American Psychiatric Publishing; 2013

DOCUMENTS (1):
  • Study Protocol (2025-05-20): https://cdn.clinicaltrials.gov/large-docs/56/NCT07098156/Prot_000.pdf